CLINICAL TRIAL: NCT01902953
Title: Prospective, Open-Label, Ex Vivo Comparison Study of Lymphoseek® and Vital Blue Dye (VBD) as Lymphoid Tissue Targeting Agents in Colon Cancer(CNC) Patients' Excised Colon w/ Abdominal Lymphatic Bed
Brief Title: Lymphoseek® as Lymphoid Tissue Targeting Agents in Colon Cancer(CNC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Danny A Sherwinter, Attending, Surgery, Maimonides Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-02-05
Record Dates: First submitted 2013-05-29; First posted 2013-07-18 (Estimated); Results first posted 2020-05-20 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: Sentinel lymph nodes; colon cancer; rectal cancer; immunohistochemistry
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymphoseek and VBD SLN dissection (Experimental): Ex-Vivo Lymphoseek and VBD SLN dissection
  Interventions: Drug: Lymphoseek and VBD Sln dissection

INTERVENTIONS:
Drug: Lymphoseek and VBD Sln dissection — See detailed description of study design
  Other Names: SLN dissection

SUMMARY:
45 patients undergoing a colon (large bowel/intestine)removal operation for the diagnosis of colon cancer will be included in this study. During colon operation the affected portion of the colon is removed. In addition, lymph nodes are included in the specimen and evaluated by a pathologist. Analysis of the lymph nodes in the specimen are important because this is an important aspect of determining the stage of the cancer.

Once the standard technique is used for the colon removal operation and the specimen is removed it will be injected with two drugs to help identify the lymph nodes. One is a blue dye and the other a radiotracer. The colon and ALL of the lymph nodes will then be sent for the standard pathologic evaluation. The patient themselves will never be injected with these drugs being used for research.

Following the standard lymph node evaluation, an additional pathologist at an outside research facility will further examine the lymph nodes in the specimen using more in depth techniques which are above and beyond the standard of care.

The results of all the pathologic tests will be conveyed to the surgeon of record to help in their decision making regarding further treatment.

The study hypothesis is that radiotracer will be at least as effective as blue dye in identifying the lymph nodes most likely to harbor cancer cells (sentinel nodes). Once identified, these sentinel nodes can then undergo a more in depth review leading to improved staging of colorectal cancer and more accurate treatment.

DETAILED DESCRIPTION:
This study is a single center, open-label, within patient's tissue ex vivo comparative study of Lymphoseek (Lymphoseek (Technetium Tc 99m Tilmanocept) is a radiotracer that accumulates in lymphatic tissue by binding to a mannose binding receptor that resides on the surface of dendritic cells and macrophages. Lymphoseek has a diameter of about 5 nm, which is substantially smaller than current radiolabeled agents used for targeting lymphoid tissue. Lymphoseek's small diameter permits enhanced diffusion into lymph nodes and blood capillaries, resulting in a rapid injection site clearance. Upon entry into the blood, the agent binds to receptors in the liver or is filtered by the kidney and accumulates in the bladder.)and vital blue dye (Patent Bleu V) in the detection of excised lymph nodes in patients with known cancer of the colon.

The colon segment with tumor and the anticipated involved nodal bed will be removed intact. After the surgical procedure is completed, the specimen is instantly taken to an extra table in the operating room. It is performed just after the specimen is taken out. The colonic specimen is incised longitudinally on the antimesenteric side.

Lymphatic mapping is employed on the specimen by using first injection Lymphoseek (50 µg/2 mCi) in 0.1-1.0 ml, followed in 15-30 min by 1 ml 1% blue dye, each injected subserosally and submucosally around the tumor (peritumoral sites employed) by using tuberculin syringe. After 5-7 minutes of massage with little circulatory movements on the lesion, the marking agents are moved into the lymphatic paths to the sentinel lymph nodes(SLN)in the mesentery.

By low level diathermy, sharp dissection of lymphatic path(s) to the SLN(s) may be existent.

Blue nodes shall be removed first by visual inspection. This inspection and dissection shall last not longer than 20 minutes. Each blue node will then be assessed for counts as well as color and the "hot" rule (3σ) applied as described below.

Following blue node removal, each sentinel lymph node can be removed from the basin and marked before the specimen is submitted for pathologic appraisal.

The Lymphoseek-designated (localized) lymph nodes are defined as lymph nodes that have a gamma detector count greater than the sum of 3 square roots of the mean background count (i.e., standard deviation) added to the mean background count. This is referred to hereafter as the "3σ rule" and as the "threshold criteria". If the gamma detector used cannot obtain gamma counts in three 2-second intervals, then one 10-second count may be used to detect gamma counts. Any lymph node count not meeting this threshold criterion will be considered a negative (non-localized) finding. The background count may be obtained by taking the 2-second counts or the 10 second counts with the handheld gamma probe extended at least 100 cm away from the injection site and the probe pointed away from anyLymphoseek source (syringes, injection site, isotope-contaminated materials).

Probing of the area will be complete when all selected node counts are negative by use of the threshold criteria. The surgeon will continue with visualization and palpation according to local practice to ensure that no grossly positive lymph nodes remain at the site of resection. To confirm the in vivo procedure, assessment of presence of a blue hue and a set of three 2-second counts or one 10-second count will be recorded for the excised lymph nodes. The mean count of the ex vivo lymph nodes will be compared to the mean of room background counts, and the same threshold criteria used to determine a positive finding for the in vivo nodes will be applied to the ex vivo specimens.

All removed lymph nodes will be sent to pathology for further evaluation. All lymph nodes will undergo enhanced pathological evaluation including serial sectioning with H&E staining as well as immunohistochemical (IHC) markers A- The primary objective of efficacy is the concordance of in vivo detection rates of Lymphoseek and VBD in excised lymph nodes as tissue phenotype is confirmed by histology.

B- The primary objective is the assessment of the excised lymph node(s) to confirm the presence/absence of tumor metastases in all nodes and a contrast of pathology findings in per agent-found nodes versus all non-agent-based removed nodes.

Secondary evaluations will include localization rates (identification of any hot and/or blue node), degree of localization (node number/patient's ex vivo total tissue), counts localized per node, and time to localization and stabilization.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided written informed consent with Health Insurance Portability and Accountability Act (HIPAA) authorization.
* The patient has a diagnosis of colon cancer and is a candidate for surgical intervention, with ex vivo lymph node mapping being a part of the surgical plan.
* The patient is at least 18 years of age at the time of consent.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of Grade 0 - 2.
* The patient has a clinical negative node status at the time of study entry (i.e., Tis-4, N0, M0).

Exclusion Criteria:

* The patient has clinical or radiological evidence of metastatic cancer including palpably abnormal or enlarged lymph nodes.
* The patient has undergone node basin surgery of any type or radiation to the nodal basin(s).
* The patient has undergone radiation therapy or chemotherapy treatment within the previous 45 days.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny A Sherwinter, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lymphoseek and VBD SLN Dissection
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lymphoseek and VBD SLN Dissection
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.94 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Lymphoseek for Detection of Sentinel Nodes
Description: Number of Participants in Concordance of in vivo detection rates of Lymphoseek and VBD in excised lymph nodes as tissue phenotype is confirmed by histology.
Time Frame: 0-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphoseek and VBD SLN Dissection
Number analyzed (Participants) | 16
Participants | 16

2. Secondary Outcome: Localization Rates
Description: Number of Participants with secondary evaluations will include localization rates (identification of any hot and/or blue node),
Time Frame: On the day of surgery i.e. day 0 of index operation
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphoseek and VBD SLN Dissection
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Arm/Group | Lymphoseek and VBD SLN Dissection
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-01): https://cdn.clinicaltrials.gov/large-docs/53/NCT01902953/Prot_SAP_000.pdf